CLINICAL TRIAL: NCT00221286
Title: Pegylated Interferon Alfa-2a Versus Emtricitabine / Tenofovir +/- Pegylated Interferon Alfa-2a for the Treatment of Chronic HBe-Ag Positive Hepatitis B Infection in HIV-Coinfected Patients - the PEGPLUS Trial
Brief Title: Efficacy and Safety of PegIFN +/- FTC / TDF to Treat Chronic Hepatitis B in HIV-Coinfected Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University Hospital, Bonn (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Prof. Jürgen K. Rockstroh, Bonn University, Germany
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ML-18150
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Hepatitis B; HIV Infections
Keywords: chronic hepatitis B; human immunodeficiency virus; pegylated interferon; tenofovir DF; emtricitabine
MeSH Terms: conditions — Hepatitis B, Chronic; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — peginterferon alfa-2a; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pegylated interferon alfa-2a
Drug: tenofovir DF / emtricitabine combination therapy
Drug: pegIFN / TDF / FTC combination therapy

SUMMARY:
The efficacy of pegylated interferons in the treatment of chronic hepatitis B has shown superior results to standard of care in patients only infected with hepatitis B. The efficacy of pegylated interferon for the treatment of chronic hepatitis B in HIV-coinfected patients is not known at present.

The purpose of this study is to evaluate the efficacy of pegylated interferon in the treatment of chronic hepatitis B in HIV-infected individuals.

Apart from evaluating the efficacy of pegylated interferon therapy in this setting as such, i.e. in patients without present or future need of highly active antiretroviral therapy (HAART) for HIV-infection, there is a second purpose of this study, to investigate whether combination treatment of HBV-infection may be superior to pegylated interferon therapy alone.

Therefore patients without need of HAART are offered pegylated interferon alfa-2a over 48 weeks. Patients who require HAART are offered emtricitabine / tenofovir DF containing HAART over 72 weeks PLUS pegylated interferon alfa-2a over 48 weeks vs. emtricitabine / tenofovir DF containing HAART over 72 weeks WITHOUT pegylated interferon-alfa-2a.

DETAILED DESCRIPTION:
Even though the generated data on standard interferon for the treatment of chronic HBV-infection in HIV-coinfected patients appears not promising at the moment, it is however the only treatment with a curative intention. Trials with pegylated interferon in the treatment of chronic HBV-infection in monoinfected patients with pegylated interferons showed higher efficacy than standard of care and when compared to historic data higher efficacy compared to non-pegylated interferon. This suggests in parallel a higher efficacy in the treatment of chronic hepatitis B in HIV-coinfected as well. At the same time, analysis suggested a further benefit when pegylated interferon therapy was prolonged beyond 24 weeks to 48 weeks as the elimination of HBV-DNA from serum appeared to continue beyond 24 weeks. Looking again at data from chronic hepatitis C infection, it is well known that the elimination kinetics of HCV-RNA in HIV-coinfected patients is slower compared to HCV-monoinfected patients, clearly suggesting rationale to offer 48 weeks pegylated interferon for the treatment of chronic hepatitis B to HIV-coinfected patients as well.

Parallel to the above said there are several other factors suggesting a positive effect of a combination treatment with nucleoside / nucleotide analogues active against HBV and interferon. Therefore patients in need for antiretroviral therapy with CD4-cells above 200/µl will be randomized to either PegIFN as part of a combination treatment with FTC and TDF or to FTC / TDF combination therapy alone. Patients receiving HAART will also receive a third active antiretroviral HIV-drug, either a non-nucleoside analogue (NNRTI) or a protease inhibitor (PI), at the choice of the investigator. A non-divergent antiretroviral therapy solely based on nucleoside analogues will not be allowed in this trial.

The objective of this study is to assess the efficacy (HBV-DNA < 5x10³ copies/ml, loss of HBe-Ag, HBe-seroconversion) and safety (adverse events, serious adverse events) of PegIFN for 48 weeks, to that of PegIFN for 48 weeks plus TDF and FTC containing HAART, to that of TDF and FTC containing HAART for 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic hepatitis B infection (> 6 months) with detectable HBV DNA > 5x100000 copies/ml (PCR-Assay) on two separate occasions
* HBe-Ag positive, anti-HBe negative
* HBs-Ag positive, anti-HBs negative
* a liver biopsy within the last 12 months prior to screening consistent with chronic hepatitis B
* Documented HIV-infection
* CD4-cell count > 200 cells/µl
* Elevated serum ALT > ULN but £ 10X ULN as determined by two abnormal values taken >14 days apart during the six months before the first dose of study drug with at least one of the determinations obtained during the screening period
* Serum-creatinine clearance > 70 ml/min, according to Cockcroft-Gault
* Anorganic phosphate > 0,65 mmol/l (2,0 mg/dl)
* Neutrophils above 1.5 G/l, Hb above 11.5 g/dl (females) or 12.5 g/dl(males), thrombocytes above 90 G/l
* Ability to understand and sign a written consent form

Exclusion Criteria:

* Older than 65 years of age, younger than 18 years of age
* Pregnancy, lactating women
* Concomitant / prior medication / hypersensitivity to study medication
* Prior use of antiretroviral therapy in particular adefovir dipivoxil, tenofovir DF, lamivudine, emtricitabine, or interferon
* Treatment with interleukin 2 or corticosteroids less than 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* Currently receiving investigational agents unless approved by the study coordinator
* History of having received any systemic anti-neoplastic (including radiation < 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study.
* Patients not receiving HAART (Arm A) must be expected not be in need for antiretroviral therapy for HIV-infection at any time during the study 72 weeks, as judged by the investigator.
* Hypersensitivity to any of the components of the study drugs (tenofovir, emtricitabine, pegylated interferon alfa-2a)

Concurrent liver disease:

* Ongoing hepatitis A, C or Delta infection: positive testing for anti HAV-IgM, HCV-RNA, anti-HDV, HDV-Ag
* Ongoing EBV or CMV infection: positive testing for anti EBV-IgM, CMV-eAg
* Autoimmune hepatitis
* Patients with a value of alpha-fetoprotein >100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months and magnetic resonance tomography of the liver shows no evidence of hepatocellular carcinoma.
* Liver cirrhosis, CHILD-Pugh Score B or C; history or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* History or other evidence of a medical condition associated with chronic liver disease other than HBV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver diseases including Wilson's and alpha1-antitrypsin deficiency, alcoholic liver disease, toxin exposures, thalassemia).
* Alcohol abuse (> 30g ethanol/d for males, > 20 g ethanol/d for females) or use of other recreational drug substances)
* Serum total bilirubin above twice the upper limit of normal
* ALT > 10 times the upper limit of normal

Neurological / psychiatric disorders:

* History of severe psychiatric conditions(ICD F30 - 33), graded by the consulting psychiatrist, in particular severe depression. Severe psychiatric disease is defined as major depression or psychosis, a period of treatment with an antidepressant medication or tranquilizer at therapeutic doses for depression or psychosis for at least 3 months, a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.
* History of a severe seizure disorder or current anticonvulsant use.

Cardiovascular disorders:

* History or other evidence of chronic pulmonary disease associated with functional limitation.
* Severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases).

Immunological disorders:

* Elevated auto-antibody findings
* History of immunologically mediated disease (e.g. inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis).
* Thyroid disease with thyroid function poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone or T4 concentrations, with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded.

Other:

* Gastrointestinal malabsorption
* Evidence of an active or suspected cancer or a history of malignancy where the risk of recurrence is ³20% within 2 years. Patients with a lesion suspicious of hepatic malignancy on a screening imaging study will only be eligible if the likelihood of carcinoma is £10% following an appropriate evaluation.
* History of organ transplantation
* History or other evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: HBeAg seroconversion (HBeAg loss and presence of anti HBe) ; intent to treat analysis. | week 48 and 72
Safety: study discontinuation due to adverse events; intent to treat analysis. | week 48

SECONDARY OUTCOMES:
Efficacy: loss of HBe-Ag,HBV-DNA < 5x10³ copies/ml(COBAS TaqMan HBV Test),decrease of HBV-DNA > 2xlog10 compared to baseline | week 48 and 72
normalization of ALT,intent to treat and as treated analysis; Viral kinetics of HBV-DNA; Paired liver biopsy comparison according to METAVIR-activity and fibrosis score. | week 48 and 72
for Arm B (B1 and B2): HIV-RNA < 50 copies/ml and CD4-cell increase intent to treat and as treated analysis | Weeks 4, 12, 24, 48 and 72
Safety: number of adverse events, according to type and severity. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen K Rockstroh, MD, PhD, Study Director — Bonn University, Germany; Martin - Vogel, MD, Principal Investigator — Bonn University
Locations (5):
- Germany (5):
  - ifi Institut für Interdisziplinäre Medizin, Hamburg, Hamburg
  - Praxis St. Georg, Hamburg, Hamburg
  - Abteilung Klinische Immunologie Zentrum Innere Medizin der Medizinischen Hochschule Hannover, Hanover, Lower Saxony
  - Immunologische Ambulanz, Medizinische Klinik und Poliklinik I, Bonn University, Bonn, North-Rhine Westfalia
  - Praxiszentrum Kaiserdamm, Berlin, State of Berlin